CLINICAL TRIAL: NCT02069951
Title: A Randomised Educational Trial of Practicing One Versus Two Laparoscopic Procedural Modules in Simulator Training for Novices on Procedure-to-procedure Transferability
Brief Title: Procedure-to-procedure Transfer Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Flemming Bjerrum, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 102169
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Surgery
Keywords: Laparoscopy; Training; Simulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Practice two procedures on a simulator (Experimental): All participants start by practicing a series of six basic skills modules until they reach a predefined proficiency level for each module. For all of the basic skills exercises proficiency is reached when the participants have passed the proficiency level for all exercises.
  Participants randomised to the intervention group will practice two procedures on a simulator. First a procedural module A (a laparoscopic appendectomy) to a predefined proficiency level. Upon reaching proficiency for procedural module A the participants will practice procedural module B (a laparoscopic salpingectomy) to a predefined proficiency level.
  Interventions: Other: Practice a procedural module on a simulator
- Practice one procedure on a simulator (No Intervention): All participants start by practicing a series of six basic skills modules until they reach a predefined proficiency level for each module. For all of the basic skills exercises proficiency is reached when the participants have passed the proficiency level for all exercises. Each exercise has to be passed twice within five consecutive attempts.
  Participants randomised to the control group will practice procedural module B (a laparoscopic salpingectomy) to a predefined proficiency level.

INTERVENTIONS:
Other: Practice a procedural module on a simulator
  Arms: Practice two procedures on a simulator

SUMMARY:
Surgical training programs using virtual reality simulators often only use basic skills training and the use of procedural training is very limited. Procedural training differs from basic skills training by requiring integration of isolated skills and decision making and planning components. However, it is unknown if it is necessary to practice all procedures before operating on actual patients or whether it is simply a matter of learning psychomotor skills and if these skills are transferable between different tasks.

The main hypothesis is that practicing a laparoscopic procedure on a simulator makes it easier to reach proficiency on a different laparoscopic procedure on the simulator because participants have already practiced the integration of isolated skills.

ELIGIBILITY:
Inclusion Criteria:

* Medical students enrolled at The Faculty of Health Science, University of Copenhagen.
* Obtained the bachelor degree in medicine.
* Signed informed consent.

Exclusion Criteria:

* Previous participation in trials involving laparoscopic training.
* Experience with laparoscopy surgery (having performed minimum one laparoscopic procedure as primary surgeon, including supervised procedures).
* No informed consent.
* Does not speak Danish on a conversational level.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The number of repetitions needed to reach a predefined proficiency level for a procedural module on a simulator | Up to 26 weeks
  The number of repetitions needed to reach a predefined proficiency level for a procedural module (a laparoscopic salpingectomy) on the simulator.

SECONDARY OUTCOMES:
The effective training time on the simulator (minutes) needed to reach the predefined proficiency level for a procedural module. | Up to 26 weeks
  The effective training time on the simulator (minutes) needed to reach a predefined proficiency level for a procedural module (a laparoscopic salpingectomy) on the simulator.

OTHER OUTCOMES:
Subjective Mental Effort Question score after the 1st repetition | Up to 26 weeks
  To score the level of stress, all the participants will be required to the Subjective Mental Effort Questionnaire after the first repetition of a procedural module. The SMEQ is a cognitive workload questionnaire with a scale of 0 to 150 points
Motor skills performance parameters | Up to 26 weeks
  1. The total path length (cumulative distance tip movement for both the right and left instrument) for the first attempt on procedural module B will be compared for the intervention and the control group.
  2. The total angular path (cumulative angular degrees for both the right and left instrument) for the first attempt on procedural module B will be compared for the intervention and the control group.
  3. The total procedure time for the first attempt on procedural module B will be compared for the intervention and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bjerrum, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Bjerrum F, Sorensen JL, Konge L, Rosthoj S, Lindschou J, Ottesen B, Strandbygaard J. Randomized trial to examine procedure-to-procedure transfer in laparoscopic simulator training. Br J Surg. 2016 Jan;103(1):44-50. doi: 10.1002/bjs.9966. Epub 2015 Oct 29. PMID 26511775
- [Derived] Bjerrum F, Sorensen JL, Konge L, Lindschou J, Rosthoj S, Ottesen B, Strandbygaard J. Procedural specificity in laparoscopic simulator training: protocol for a randomised educational superiority trial. BMC Med Educ. 2014 Oct 10;14:215. doi: 10.1186/1472-6920-14-215. PMID 25304939
- See also: JMC Simulation Unit — http://www.rigshospitalet.dk/RHenglish/Menu/Departments+and+Clinics/Juliane+Marie+Centre/Research/Simulation+unit+JMC/Simulation+Unit+JMC.htm